CLINICAL TRIAL: NCT03763578
Title: Licorice Versus Standard Preventive Measures for the Prevention of Caries Incidence in Young Egyptian Adults: Randomized Controlled Trial
Brief Title: Dental Caries Prevention by a Natural Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Ahmed Mady, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18941
Record Dates: First submitted 2018-11-10; First posted 2018-12-04 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Licorice (Experimental): licorice is one of the natural products that is listed by the Food and Drug Administration (FDA) as GRAS (generally regarded as safe) when used as food flavoring and sweetening agent which has an antimicrobial, anti-inflammatory and antiviral activity.
  Interventions: Other: Licorice
- Chlorhexidine (Active Comparator): The "gold standard" of oral therapeutics is Chlorhexidine due to its prolonged broad- spectrum antimicrobial effect.
  Interventions: Other: Licorice
- Control Group (No Intervention): Participants in this group will follow only the standard preventive measures which is brushing twice a day after breakfast and before bed time and daily flossing interdentally before bed time. (No Mouthwash is used)

INTERVENTIONS:
Other: Licorice — Natural herbal product
  Other Names: Glycyrrhiza glabra Linn; Mulethi
  Arms: Chlorhexidine; Licorice

SUMMARY:
The objective is to conduct an RCT to evaluate the effectiveness of Licorice in comparison to standard caries preventive measures for the prevention of new carious lesions in high caries risk patients.

DETAILED DESCRIPTION:
Research hypothesis (Null hypothesis):

The present clinical trial will be conducted to reject or accept the null hypothesis that using Licorice extract mouth wash in addition to standard preventive measures will not differ from using standard preventive measures alone in preventing incidence of new carious lesions.

PICOTS:

P: Population with high caries risk patients

I: Use of licorice.

I2: Use of chlorhexidine

C: Use of standard preventive measures (tooth brushing, tooth paste, interdental cleaning).

O.1: Primary outcome is incidence of new carious lesions

T: Time for measurement is 12 months

S: A Randomized controlled clinical trial (Parallel study)

ELIGIBILITY:
Inclusion Criteria:

* Patients with high caries risk,
* 18-25 years,
* Males or females,
* Medically free patients,
* Patients approving to participate in the study.

Exclusion Criteria:

* Patients who were on antibiotic therapy or corticosteroid therapy for 30 days before the examination,
* Patients had history of professional cleaning in the last 15 days,
* Patients with exposed pulp,
* Evidence of parafunctional habits,
* Patients with developmental dental anomalies,
* Patients undergoing or will start orthodontic treatment,
* Patients with removable prosthesis,
* Periapical Abscess or Fistula.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of new carious lesions | 12 months
  Appearance of new carious lesions within the study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Conservative and Esthetic Dentistry Department-Faculty of Dentistry- Cairo University, Cairo, Choose Any State/Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided